CLINICAL TRIAL: NCT04389190
Title: Radiation Dose Reduction Using Advanced Fluoroscopy Options in Coronary Cath Lab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tabba Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Radiation Dose Reduction trial
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Radiation Exposure; Coronary Artery Disease
Keywords: Radiation exposure, Cardiac cath lab, radiation dose monitoring
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This will be a single center non blinded quasi experimental design. Data will be collected prospectively.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Protocol (Active Comparator): This is the fluoroscopy protocol used routinely in most catheterization labs in the region. This includes fluoroscopy and cine image acquisition at 15 frames per second (FPS) at 8-inch mode. Virtual collimation and last image hold (LIH) will be used as needed. This protocol will be implemented for 6 weeks.
  Interventions: Other: Fluoroscopy settings for image acquisition
- Low frame rate protocol (Experimental): This will have fluoroscopy and cine image acquisition at 7.5 FPS at 8-inch mode with all other settings on factory default. Virtual collimation and LIH will be used as needed. This protocol will be implemented for 6 weeks as well.
  Interventions: Other: Fluoroscopy settings for image acquisition
- Customized Protocol (Experimental): This will have varying settings based on three weight based groups. Small (<60 kg), medium (60-85 kg), large (>85 kg). The variables changed are fluoroscopy dose per frame, fluoroscopy frame rate, image acquisition frame rate, thickness of the spectral beam filters, peak tube voltage and peak cathode current. Additional features will also be utilized including live zoom (1.4 factors with 12 inch field of view, FOV), fluoro store and Spot fluoroscopy. Virtual collimation and LIH will be used as needed. This protocol will be applied for 12 weeks.
  Interventions: Other: Fluoroscopy settings for image acquisition

INTERVENTIONS:
Other: Fluoroscopy settings for image acquisition — X-ray radiation is routinely used for imaging in coronary cath labs. Intervention involves lowering patient and operators X-ray exposure by employing various setting on the fluoroscopy machine.
  Other Names: Fluoroscopy settings on Infinix i8000V, Toshiba America Medical Systems, Inc

SUMMARY:
Fluoroscopy is integral part of diagnostic and therapeutic cardiac procedures. Among medical personnel, interventional cardiologists have the highest per head per year exposure to ionizing radiation which is two to three times greater than the radiologists. Although the patients' exposure is well below the level associated with increased cancer risk, yet as mentioned above, any exposure can be harmful and must be minimized using all possible dose reduction methods under the principle of 'As Low as Reasonably Achievable' (ALARA).

Radiation exposure is influenced by factors that are dependent on patient (weight, body habitus), procedure (access site, procedure complexity, use of protective shielding, collimation) and equipment (overall quality control, field of view, beam filters thickness, pulse rate etc.). In fact in modern fluoroscopic equipment, several settings are customizable to aid reduce total emitted X-ray dose. In a diverse coronary lab as Tabba Heart institute, in addition to training the lab staff on reducing radiation exposure and use of protective gear, employment of a modern X ray system Like Toshiba (Infinix i8000V, Toshiba America Medical Systems, Inc.); equipped with customizable radiation dose reduction technologies and DTS, provides the interventionists an essential tools to ensure the highest radiation safety standards. Data is still scanty to show the difference in patients and operators' radiation exposures by using tailored equipment settings. We aim to apply customized fluoroscopy protocols based on low fps and other customizable settings (thickness of the spectral beam filters, peak tube voltage and peak cathode current, live zoom (1.4 factors with 12 inch FOV), fluoro store and Spot fluoroscopy) and then assess if they significantly affect the radiation exposure of the patient and the interventionist.

DETAILED DESCRIPTION:
Fluoroscopy is integral part of diagnostic and therapeutic cardiac procedures. Due to the ionizing effect of X-rays; patients, interventionist and cath lab staff are at risk of radiation hazards that are broadly divided into two categories. One is deterministic; where severity of the injury to the exposed area is dose dependent and there is a safety threshold; the other is stochastic or probabilistic where any radiation dose can cause genetic mutation and cancers and no dose is considered safe. Among medical personnel, interventional cardiologists have the highest per head per year exposure to ionizing radiation which is two to three times greater than the radiologists. Although the patients' exposure is well below the level associated with increased cancer risk, yet as mentioned above, any exposure can be harmful and must be minimized using all possible dose reduction methods under the principle of 'As Low as Reasonably Achievable' (ALARA).

Radiation exposure is influenced by factors that are dependent on patient (weight, body habitus), procedure (access site, procedure complexity, use of protective shielding, collimation) and equipment (overall quality control, field of view, beam filters thickness, pulse rate etc.). In fact in modern fluoroscopic equipment, several settings are customizable to aid reduce total emitted X-ray dose. A lower frame rate of 7.5 frames per second (fps) compared with standard 15fps substantially reduces X-ray exposure (30% relative exposure reduction in operator dose and 19% in patient dose) without compromise in image quality. Using live zoom to digitally enlarge images also lowers the dose by 40-50% (1.4 factors with 6 inch field of view). Another significant advancement is 'Dose Tracking System' (DTS) which calculates the precise radiation dose to the patient's skin and displays the cumulative dose values as a color map on a patient graphic for immediate feedback to the interventionist. This knowledge of the exposure in real time too helps physicians adjust their practices accordingly.

In a diverse coronary lab as Tabba Heart institute, in addition to training the lab staff on reducing radiation exposure and use of protective gear, employment of a modern X ray system Like Toshiba (Infinix i8000V, Toshiba America Medical Systems, Inc.); equipped with customizable radiation dose reduction technologies and DTS, provides the interventionists an essential tools to ensure the highest radiation safety standards. Data is still scanty to show the difference in patients and operators' radiation exposures by using tailored equipment settings. We aim to apply customized fluoroscopy protocols based on low fps and other customizable settings (thickness of the spectral beam filters, peak tube voltage and peak cathode current, live zoom (1.4 factors with 12 inch FOV), fluoro store and Spot fluoroscopy) and then assess if they significantly affect the radiation exposure of the patient and the interventionist.

AIMS/OBJECTIVES

1. To compare the effect of three different fluoroscopy protocols on patient and operator's total X ray dose in coronary catheterization lab at Tabba Heart Institute, Karachi.
2. To assess the effect of low frames per seconds settings in cine imaging and fluoroscopy on quality of image during coronary procedures METHODS

Study Design:

This will be a single center non blinded quasi experimental design. Data will be collected prospectively. Study population includes patients coming for coronary procedures to the cath lab equipped with Toshiba America Medical Systems Inc., Infinix i8000V with Dose Tracking System (DTS).

Setting: Cardiac cath lab (CCL) of Tabba Heart Institute Karachi, Pakistan, (THI).

Tabba heart institute is a 160 bedded cardiac tertiary care hospital with 24 hrs emergency and facilities for primary PCI and cardiac surgeries. The institution has two fully equipped cardiac catheter labs. There is a fully trained and experienced faculty of more than 15 cardiologists and 06 interventional. On average in THI we perform diagnostic angiograms and slightly more than 1400 PCIs per year, 20% of which are for STEMI patients. This is one of the major referral centers in the city for primary PCI. THI is also a teaching hospital with approved training programs in adult cardiology and interventional cardiology.

Duration of study: Six months (24 weeks) We plan to start patient recruitment in June 2020 contingent on approval from the Ethical Review Committee. Since our monthly numbers in the cath lab exceed 200 (diagnostic angiogram and interventional procedures) each month and this is a 24/7 active cath lab with facility for primary PCI, at least six months will be ample time to meet the sample size.

Non probability sampling will be done to enroll patients in CCL. Consecutive patients presenting at CCL of THI will be assessed for eligibility. We plan to implement the three protocols weekly basis to avoid protocol implementation errors during after-hours. The weeks will be designated in a way that the customized protocol will be implemented on alternate weeks and during rest of the weeks; standard and low FPS protocol will be implemented randomly thus resulting in total recruitment period of twelve weeks for customized approach and six weeks each for the other two arms. The machine settings will be adjusted every week same time on Monday morning for the next seven days. All the patients coming to CCL during the seven days will have their procedures performed on the designated fluoroscopy protocol for that week. At the end of each week; protocol will be switched to one of the other intervention protocols. The operators will be un-blinded to the current protocol on the machine however DTS based Real time exposure will be kept hidden during the trial except for the last 3 weeks of the customized protocol.

Old calculation: For 03 pairwise comparisons, to detect significant difference among mean air Kerma (adjusted mean total x-ray dose) as a measure of patient's exposure, Mean and standard deviation used for the study were derived from (ref). We anticipated 20% reduction in radiation exposure between the standard and reduced FPS groups and 30% reduction between standard and customized protocol.

With alpha of 5% and power of 80%, sampling ratio of 1:1:2 for standards: reduced FPS: customized protocol respectively, total sample size needed is 404 with 101 patients in first two groups and 202 in customized group. To account for sampling errors and incomplete information and to maintain post hoc power, 120 patients will be included in first two groups and 240 in customized protocol. The final sample size will be 480 patients.

COVARIATES:

The covariates will include age in years, gender, height, weight, presence of major cardiac co-morbid conditions [diabetes mellitus (DM), hypertension (HTN), dyslipidemia, smoking, family history of premature coronary artery disease (CAD)] will be recorded. Indication (ACS vs. No ACS) and timing of procedure (elective, emergent, urgent) will be recorded. Type of procedure (CAG only, PCI only, combined CAG and PCI), Native versus graft angiogram, LV gram performed as part of the study will also be documented. Procedure details including number of operators, type of operator (fellow/faculty), access sites (femoral/radial), procedure duration, and contrast volume will be recorded. . In case of PCI, single or multi vessel PCI, number of vessels treated, numbers and sizes of stents and catheters used, PCI complexity, (High B/C or Non High B/C), bifurcation lesion and graft angioplasty will be documented. Variables related to radiation dose reduction: fluoro duration in minutes, number of cine and/or fluoro stores, fluoroscopy dose per frame, fluoroscopy frame rate, image acquisition frame rate, thickness of the spectral beam filters, peak tube voltage and peak cathode current will be recorded. The customized settings on these variables vary according to patient's weight and will be stratified accordingly. Use of live zoom and spot fluoro will also be recorded. Outcome variables include patient's exposure (air kerma (Gy), dose area product (DAP) (Gy/cm2) and peak skin dose (PSD) in mGy) and operators' exposure (μSv).

PLAN OF STATISTICAL ANALYSIS Primary analysis: Means ± SD will be reported for continuous variables if normally distributed (confirmed by constructing Histograms, Shapiro-Wilk's W tests and normal probability plots) or median ±IQR if not normally distributed. Percentages will be used for categorical variables.

For primary outcome of patient and operator X-ray dose, Independent sample t-test or Man Whitney U test will be used, depending about distribution of the variables, for comparison of two individual fluoroscopy protocols. One way ANOVA will be used for multiple comparisons of the three protocols and for post hoc correction Bonferroni test will be utilized. Tukey's HSD will be used for comparison of individual means. Results will be stratified according to the type of procedure (Diagnostic angiogram vs. PCI). Univariate analysis will be performed to assess important predictors of radiation dose of operator and patients. Multivariable linear regression analysis will be performed for adjustment of important confounding variables.

Secondary analysis: For secondary analysis on quality of images, Kruskal Wallis analysis of ranks test will be employed for multiple group comparisons.

Additional analysis: The customized approach will be further divided in three sub groups according to weight of the patients settings Primary outcomes will also be compared across these subgroups from the standard protocol.

Pearson's correlation will be used and correlation coefficients will be generated to assess the association of patient's skin dose with fluoro time, contrast volume and DAP.A P-value <0.05 will be taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* percutaneous coronary interventional (PCI) and other fluoroscopy assisted cardiac procedures including valvular interventions and device closures.
* Both emergent and elective procedures.
* Patients undergoing procedures both via trans-radial or trans-femoral approach will be included.

Exclusion Criteria:

* Intra-cardiac device insertions and procedures requiring digital subtraction angiography (DSA) will be excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
patient and operator radiation exposure | within 24 hours
  Operator dose (μSv): Exposure of X-ray to the first and second operator will be measured using the Raysafe i2 system (Unfors Raysafe, Sweden). The personal dosimeter (PDM) in this consists of semiconductors layered with a film and provides real time dose information. All operators will wear the PDM on left side on upper torso. PDM readings will be obtained on an individual procedure basis and readings will be hidden from the operators.
  Patient total X-ray dose: This will be calculated by obtaining adjusted mean total x-ray dose i.e. air kerma (Gy), dose area product (DAP) (Gy/cm2) and real time Peak skin dose in mGy using Toshiba Inc.'s dose tracking system.

SECONDARY OUTCOMES:
quality of imaging | within 24 hours
  This includes quality of imaging as assessed by the interventional cardiologists in our cath lab. This will be judged on 10 point scale where 10 means ideal image and 1 means worst image. Quality of image will be measured on basis of optimal resolution, image contrast, clarity of cardiac motion, and tertiary branch visibility. Aggregate scores will be calculated for each study based on individual images. Assessors will be blinded to the frame rate and machine settings for that study.

CONTACTS AND LOCATIONS:
Overall Officials: Asad Z Pathan, MD, Principal Investigator — Tabba Heart Institute
Locations (1):
- Tabba Heart Institute, Karachi, Sindh, Pakistan